CLINICAL TRIAL: NCT03483012
Title: A Phase II Study of Atezolizumab in Combination With Stereotactic Radiation for Patients With Triple-negative Breast Cancer and Brain Metastasis
Brief Title: Atezolizumab + Stereotactic Radiation in Triple-negative Breast Cancer and Brain Metastasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nancy Lin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-519
Record Dates: First submitted 2018-02-28; First posted 2018-03-29 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Stereotactic radiosurgery (SRS) (Experimental): * Atezolizumab administered intravenously once every 3 weeks
  * Stereotactic radiosurgery (SRS) begin within 14 days after brain MRI obtained
  Interventions: Drug: Atezolizumab; Procedure: Stereotactic radiosurgery (SRS)

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is a protein that affects your immune system by blocking the PD-L1 pathway
  Other Names: Tecentriq
Procedure: Stereotactic radiosurgery (SRS) — Stereotactic radiosurgery (SRS) is a standard procedure used to treat patients with cancer in the brain. SRS uses many precisely focused radiation beams to treat tumors

SUMMARY:
This research study is studying the combination of a drug called atezolizumab and a radiation procedure called stereotactic radiosurgery (SRS) as a possible treatment for triple-negative breast cancer that has spread to the brain.

The interventions involved in this study are:

* Atezolizumab
* Stereotactic radiosurgery (SRS)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved atezolizumab for this specific disease but it has been approved for other uses.

Atezolizumab is a protein that affects the immune system by blocking the PD-L1 pathway. The PD-L1 pathway controls the body's natural immune response, but tumors can interrupt this pathway and partially resist or escape the immune system. By blocking the PD-L1 pathway, Atezolizumab may help the immune system identify and catch tumor cells.

Stereotactic radiosurgery (SRS) is a standard procedure used to treat patients with cancer in the brain. SRS uses many precisely focused radiation beams to treat tumors. It is not surgery in the traditional sense because there's no incision. Instead, SRS uses 3-D imaging to target high doses of radiation to the affected area with minimal impact on the surrounding healthy tissue. Like other forms of radiation, SRS works by damaging the DNA of the targeted (tumor) cells. The affected cells then lose the ability to reproduce, which causes tumors to shrink.

When given separately, atezolizumab and SRS, work in different ways to help stop cancer cells from growing and spreading. However, it is not known if giving atezolizumab and SRS at the same time will have a better effect than giving each treatment on its own. It is hoped that SRS treatment will damage cancer cells and make them more visible to the immune system.

The researchers conducting this study are testing to see whether giving SRS with atezolizumab may boost the body's immune response to cancer, and therefore improve upon the effects of either SRS or atezolizumab given alone.

In this research study, the investigators will measure the length of time that the participant receive this study intervention without the disease getting worse. The investigators will also look at how well the disease responds to atezolizumab and SRS as well as the safety of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed Stage IV invasive breast cancer. Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Either the primary tumor and/or metastatic tumor must be triple-negative as defined below:

  * Hormone receptor status: the invasive tumor must be ER- and PR-negative, or staining present in <1% by immunohistochemistry (IHC)
  * HER2 status: the invasive tumor must be Human Epidermal Growth Factor Receptor 2 Negative (HER2-negative) by the ASCO CAP guidelines
* In cases where both primary tumor and metastatic sample(s) have been tested for ER, PR, and HER2, the triple-negative status of the most recent sample should be used.
* Participants must have a diagnosis of brain metastases for which SRS is indicated, as determined by a radiation oncologist.
* The contrast-enhancing intraparenchymal brain metastases(s) must be well circumscribed and must have a maximum diameter of ≤ 3.0 cm in any direction on the enhanced scan.
* Participants must not have more than 5 new or progressive lesions in the brain requiring SRS treatment (greater than 5 total brain lesions are allowed as long as no more than 5 lesions require SRS treatment).
* Participants must have measurable extracranial disease as defined by RECIST 1.1.
* Participants must be willing to undergo a research biopsy at baseline and at Cycle 2 Day 1 if extracranial metastases are safely accessible. Participants for whom biopsies cannot be safely performed must be willing to submit an archival primary and/or metastatic specimen. The biopsies may be waived with prior PI approval for the first 6 participants enrolled to the safety run in phase.
* Prior systemic therapy:

  * Participants must have discontinued systemic therapy at least 14 days prior to initiating protocol therapy.
  * There is no limit to the number of prior lines of systemic therapy. Participants who have not received any systemic therapy for metastatic disease are also eligible.
  * Participants may initiate or continue bisphosphonate therapy on study.
* Prior local therapy:
* Prior surgery, whole brain radiation or SRS is allowed as long as the most recent brain progression is amenable to SRS treatment.
* Resolution of all chemotherapy-related or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (≤ Grade 2 allowed) and alopecia (of any grade).
* Participant is ≥18 years old.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Stable dose of dexamethasone 2mg or less for at least 7 days prior to initiation of treatment
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/μl
  * platelets ≥75,000/μl
  * hemoglobin ≥9 g/dL
  * total bilirubin ≤1.5mg/dL (≤2.0 in patients with known Gilberts syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN. ≤5.0 × institutional ULN for patients with documented liver metastases.
  * albumin >2.5mg/dL
  * serum creatinine ≤1.5mg/dL or calculated GFR ≥60 mL/min
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 8 days of initiating protocol therapy.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of study treatment. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. The effects of atezolizumab on the developing human fetus are unknown and radiotherapy has known teratogenic effects so women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 4 months after completion of atezolizumab administration.
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document

Exclusion Criteria:

* CNS complications for whom urgent neurosurgical intervention is indicated (e.g., resection, shunt placement).
* Known leptomeningeal or brainstem metastases. The presence of leptomeningeal enhancement alone, without associated clinical manifestations and/or positive CSF cytology, will not be constituted as known leptomeningeal metastases.
* Treatment with high dose systemic corticosteroids defined as dexamethasone >2mg/day or bioequivalent within 7 days of initiating therapy.
* Patients unable to undergo gadolinium contrast-enhanced MRI or receive IV contrast for any reason (e.g., due to pacemaker, ferromagnetic implants, claustrophobia, extreme obesity, hypersensitity).
* Participants who are receiving any other investigational agents.
* Previous treatment with any anti-PD-1, PD-L1, or PD-L2 agent.
* Subjects with a history of hypersensitivity to compounds of similar biologic composition to atezolizumab or any constituent of the product
* The participant has an uncontrolled intercurrent illness, including, but not limited to uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure-New York Heart Association Class III or IV, active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus, gastric or duodenal ulceration diagnosed within the previous 6 months, severe malnutrition or psychiatric illness/social situations that would limit compliance with study requirements.
* Participant has a medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication. For example, patients with autoimmune disease that requires systemic steroids or immunosuppression agents should be excluded. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has evidence of active, noninfectious pneumonitis that requires treatment with steroids.
* Has a history of interstitial lung disease.
* The participant is known to be positive for the human immunodeficiency virus (HIV), HepBsAg, or HCV RNA. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with atezolizumab.
* Individuals with a history of different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the principal investigator to be at low risk for recurrence of that malignancy.
* Has received a live vaccine within 28 days of planned start of study therapy.
* The participant is pregnant or breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy U Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab + Stereotactic Radiosurgery (SRS): * Atezolizumab administered intravenously once every 3 weeks
  * Stereotactic radiosurgery (SRS) begin within 14 days after brain MRI obtained
  Atezolizumab: Atezolizumab is a protein that affects your immune system by blocking the PD-L1 pathway
  Stereotactic radiosurgery (SRS): Stereotactic radiosurgery (SRS) is a standard procedure used to treat patients with cancer in the brain. SRS uses many precisely focused radiation beams to treat tumors
Period: Overall Study
Arm/Group | Atezolizumab + Stereotactic Radiosurgery (SRS)
Started | 6
Completed | 0
Not Completed | 6
Not completed — Lack of Efficacy | 6

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 46 [32 to 69]
Age, Customized [Count of Participants; unit: Participants]
  Age category: <50 | 4
  Age category: >=50 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants]
  0-Fully active, able to carry on pre-disease performance without restriction | 5
  1-Restricted in strenuous physical activity but able to perform work of a light or sedentary nature | 1
Stage at initial diagnosis [Count of Participants; unit: Participants]
  I- Cancer has spread to other tissue in small area | 1
  II- Tumor is 20-50mm with some lymph node involvement, or tumor is >50mm with no nodal involvement | 4
  Not IV but otherwise unknown- Non-metastatic but stage otherwise unknown | 1
Disease-free interval (interval from primary diagnosis date to metastatic diagnosis date) [Count of Participants; unit: Participants]
  <2 years | 2
  >=2 years | 4
Hormone receptor status of primary tumor [Count of Participants; unit: Participants]
  ER positive/PR negative | 1
  ER and PR negative | 5
Hormone receptor status of metastatic tumor [Count of Participants; unit: Participants]
  ER and PR negative | 1
  Not done | 5
HER-2 status of primary tumor (IHC) [Count of Participants; unit: Participants]
  Negative (0,1+) | 4
  Equivocal (2+) | 1
  Not done | 1
HER-2 status of primary tumor (ISH) [Count of Participants; unit: Participants]
  Negative (copy number <4 and HER2/CEP17 ratio <2.0) | 4
  Not done | 2
Measurable disease by RECIST 1.1 at baseline [Count of Participants; unit: Participants]
  Yes | 5
  No | 1
Prior adjuvant or neoadjuvant endocrine therapy [Count of Participants; unit: Participants]
  Yes | 3
  No | 3
Prior lines of chemotherapy for metastasis or recurrence [Count of Participants; unit: Participants]
  0 lines | 2
  1 line | 3
  >=2 lines | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Defined as time from first dose of atezolizumab (day 1 cycle 1) to progression or death due to any cause. Progression is defined according to the bi-compartmental model proposed in the RANO-BM publication, and is defined as the first detection of radiologic progression of intracranial (per RANO-BM criteria), extracranial (per RECIST 1.1 criteria), or both or unequivocal progression of non-measurable disease in the opinion of the treating physician; with each compartment (CNS and non-CNS) assessed separately
Time Frame: Assessed from the first dose of atezolizumab until the date of first documented progression according to RANO-BM or date of death from any cause, whichever came first, for a maximum of 1.5 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Atezolizumab + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 6
weeks | 5.8 [4.1 to NA] — Insufficient sample size/number of events

2. Secondary Outcome: Extracranial Objective Response Rate
Description: Defined as the percentage of patients achieving a complete response (complete disappearance of all target and non-target lesions; no new lesions) or partial response (at least 30% decrease in the sum of the diameters of target lesions; persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits [i.e., "non-CR/non-PD" in non-target lesions]; and no new lesions) based on RECIST 1.1
Time Frame: Assessed from the first dose of atezolizumab until disease progression, intercurrent illness, unacceptable toxicity, noncompliance/withdrawal, or general/specific worsening of condition, for a maximum of 1.5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Atezolizumab + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 6
percentage of patients | 0 [0 to 45.9]

3. Secondary Outcome: Overall Survival
Description: Defined as the time from first dose of atezolizumab (day 1 cycle 1) to death from any cause. Patients who are alive at the end of the study are censored at the date of last known alive.
Time Frame: Assessed from the first dose of atezolizumab to the date of death from any cause or date last known alive, for a maximum of 3.8 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Atezolizumab + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 6
weeks | 42.4 [15.7 to NA] — Insufficient sample size/number of events

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on the first day of each treatment cycle, at the end of treatment, and up to 30 days post-end of treatment, for up to a maximum of 1.8 years. Death events were assessed for up to a maximum of 3.8 years.
Arm/Group | Atezolizumab + Stereotactic Radiosurgery (SRS)
All-Cause Mortality (participants affected / at risk) | 5/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab + Stereotactic Radiosurgery (SRS) (N=6)
Intracranial hemorrhage (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab + Stereotactic Radiosurgery (SRS) (N=6)
Cushingoid (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Pharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT03483012/Prot_SAP_000.pdf